CLINICAL TRIAL: NCT01228903
Title: Is Uric Acid a Mediator of Endothelial Dysfunction in Patients With Chronic Kidney Disease?
Brief Title: Uric Acid and the Endothelium in CKD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 10-0625; K23DK088833 (NIH)
Record Dates: First submitted 2010-10-25; First posted 2010-10-27 (Estimated); Results first posted 2017-02-23 (Actual); Last update posted 2017-06-28 (Actual); Status verified 2017-05

CONDITIONS: Kidney Disease
Keywords: uric acid kidney disease endothelial dysfunction
MeSH Terms: conditions — Kidney Diseases | interventions — Allopurinol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control (Placebo Comparator): Patients who are randomized to this group will received placebo tablets. Placebo tables do not contain an active ingredient. This group will be used as a baseline group to compare the effects of lowering uric acid on vascular function.
  Interventions: Other: Placebo
- Allopurinol (Active Comparator): Patients who are randomized to this group will receive allopurinol tablets. Allopurinol is a medicine that lowers uric acid levels. The effects of lowering uric acid on vascular function outcomes will be assessed and compared to the control group.
  Interventions: Drug: Allopurinol

INTERVENTIONS:
Drug: Allopurinol — Xanthine oxidase inhibitor- effective at lowering uric acid levels.
  Other Names: Zyloprim, Allohexal, Allosig, Milurit, Alloril, Progout, Zyloric.
  Arms: Allopurinol
Other: Placebo — Placebo tablets with no active ingredient
  Arms: Control

SUMMARY:
This study will test the hypothesis that uric acid impairs the function of vessels in patients with kidney disease

DETAILED DESCRIPTION:
The purpose of the study is to understand the effect of lowering serum uric acid levels on vascular function in individuals with chronic kidney disease by comparing the effects of:

1) Allopurinol therapy and 2) Placebo.

Patients will receive: 3 month study drug (either allopurinol or placebo), with assessment of serum uric acid levels and vascular function.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with moderate chronic kidney disease (CKD stage III) with estimated glomerular filtration rates between 30-60 mL/min/ 1.73m2
* Elevated uric acid levels
* Age range: more than 18 years old
* Ability to give informed consent
* Albumin > 3.0 g/dL
* BMI < 40 kg/m2

Exclusion Criteria:

* Life expectancy < 1.0 years
* Expected to undergo living related kidney transplant in 6 months
* Pregnant, breast feeding, or unwilling to use adequate birth control
* History of severe liver disease
* History of severe congestive heart failure
* History of hospitalizations within 3 months
* Active infection, on antibiotics
* History of Warfarin Use or other medications that are contraindicated with allopurinol
* Uncontrolled hypertension
* History of acute gout on Allopurinol
* History of adverse reaction to Allopurinol
* Immunosuppressive therapy within the last 1 yr

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2010-10; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Diana Jalal, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado at Denver, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be made available to investigators upon request from the PI

REFERENCES:
- [Derived] Perrenoud L, Kruse NT, Andrews E, You Z, Chonchol M, Wu C, Ten Eyck P, Zepeda-Orozco D, Jalal D. Uric Acid Lowering and Biomarkers of Kidney Damage in CKD Stage 3: A Post Hoc Analysis of a Randomized Clinical Trial. Kidney Med. 2020 Feb 26;2(2):155-161. doi: 10.1016/j.xkme.2019.11.007. eCollection 2020 Mar-Apr. PMID 32964203
- See also: What is the endothelium? — http://en.wikipedia.org/wiki/Endothelium

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Control | Allopurinol
Started | 41 | 39
Completed | 36 | 34
Not Completed | 5 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | Allopurinol | Total
Number analyzed (Participants) | 41 | 39 | 80
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.9 (9.3) | 55.9 (13.7) | 57.4 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 7 | 16
  Male | 32 | 32 | 64
Region of Enrollment [Number; unit: participants]
  United States | 41 | 39 | 80

OUTCOME MEASURES:

1. Primary Outcome: Change in Endothelial Dependent Dilation From Baseline to Week 12
Description: Change in Endothelial Dependent Dilation measured by Flow Mediated Dilation at baseline and week 12
Time Frame: Baseline and 12 weeks
Measure: Mean (Standard Deviation); unit: % change
Groups:
- Allopurinol: Allopurinol: Xanthine oxidase inhibitor
Arm/Group | Control | Allopurinol
Number analyzed (Participants) | 41 | 39
% change | 0.2 (4.1) | 0.9 (3.9)
Statistical Analysis 1: Comparison: Control vs Allopurinol; The null hypothesis was the there will be no difference between the placebo and allopurinol. The power for the study was calculated (as appropriate) based on the prior literature; Test type: Equivalence — (Doehner et al.) CHF patients on allopurinol (n= 14) had improved BA-FMD= 10.6 ± 2.0 (mean ± SE) vs placebo (n= 14, FMD= 6.7 ± 0.1); difference in means= 3.9. Yiginer et al. found a similar difference in metabolic syndrome. A sample size of 34/group will have 80% power to detect a difference in means of 3.9 (common standard deviation=5.6, two group t-test=0.050 two-sided significance). Accounting for a potential drop-out rate17%, n= 40/group was recruited; p = 0.47, Wilcoxon (Mann-Whitney); Mean Difference (Net) = 0.7 — The estimated value represents the difference between the change from baseline in both groups

2. Secondary Outcome: Change in C-reactive Protein From Baseline to Week 12
Time Frame: Baseline and 12 weeks
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Control | Allopurinol
Number analyzed (Participants) | 41 | 39
mg/L | 0.7 (3.4) | 00.42 (9.5)

3. Secondary Outcome: Change in Serum Interleukin-6 From Baseline to Week 12
Time Frame: Baseline and 12 weeks
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Control | Allopurinol
Number analyzed (Participants) | 41 | 39
pg/mL | 0.15 (3.1) | 0.37 (2.7)

4. Secondary Outcome: Change in Monocyte Chemotactic Protein-1 From Baseline to Week 12
Time Frame: Baseline and 12 weeks
Population: -4.7
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Control | Allopurinol
Number analyzed (Participants) | 41 | 39
pg/mL | -4.7 (45.8) | 3.6 (36.7)

5. Secondary Outcome: Change in Oxidized Low Density Lipoprotein From Baseline to Week 12
Time Frame: Baseline and 12 weeks
Measure: Mean (Standard Deviation); unit: u/L
Arm/Group | Control | Allopurinol
Number analyzed (Participants) | 41 | 39
u/L | -0.08 (11.8) | -2.97 (16.4)

6. Other Pre Specified Outcome: Change in Serum Uric Acid Levels From Baseline to Week 12
Description: Serum uric acid levels were measured both at baseline and after 12 weeks
Time Frame: Baseline and 12 weeks
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Control | Allopurinol
Number analyzed (Participants) | 41 | 39
mg/dL | 0.05 (1.54) | 3.24 (1.35)

ADVERSE EVENTS:
Arm/Group | Control | Allopurinol
Serious Adverse Events (participants affected / at risk) | 0/41 | 1/39
Other Adverse Events (participants affected / at risk) | 9/41 | 4/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control (N=41) | Allopurinol (N=39)
Death (Cardiac disorders) | 0 (0) | 1 (1) — One patient died in the allopurinol arm, and it was attributed to a cardiovascular event
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Control (N=41) | Allopurinol (N=39)
gout (Musculoskeletal and connective tissue disorders) | 1 | 1
GI discomfort (Gastrointestinal disorders) | 2 | 2
rash (Skin and subcutaneous tissue disorders) | 2 | 0
Abnormal Liver Function Tests (Hepatobiliary disorders) | 2 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No